CLINICAL TRIAL: NCT06679959
Title: A Phase I/IIa, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ASC30 Injection, for Subcutaneous Use in Participants With Obesity
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ASC30 Injection in Participants With Obesity
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC30-101
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- SAD Cohort 1 (Experimental): SAD Dose 1
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 2 (Experimental): SAD Dose 2
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 3 (Experimental): SAD Dose 3
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 4 (Experimental): SAD Dose 4
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 5 (Experimental): SAD Dose 5
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 6 (Experimental): SAD Dose 6
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 7 (Experimental): SAD Dose 7
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- SAD Cohort 8 (Experimental): SAD Dose 8
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- MAD Cohort 1 (Experimental): MAD Dose 1
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- MAD Cohort 2 (Experimental): MAD Dose 2
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo
- MAD Cohort 3 (Experimental): MAD Dose 3
  Interventions: Drug: ASC30 Injection, for subcutaneous use or placebo

INTERVENTIONS:
Drug: ASC30 Injection, for subcutaneous use or placebo — Drug: ASC30 injection, for subcutaneous use Drug: Placebo injection, for subcutaneous use

SUMMARY:
This randomized, double-blind, placebo-controlled single ascending dose (SAD)/ multiple ascending dose (MAD) study is designed to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASC30 injection

ELIGIBILITY:
Inclusion Criteria:

1. Have provided informed consent before initiation of any study-specific procedures.
2. Male or female participants, non-smokers, between 18 and 65 years of age (both inclusive).
3. No clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and other screening procedures.

Exclusion Criteria:

1. Have evidence of any clinically significant active or chronic disease.
2. Have any prior diagnosis of diabetes mellitus (T1DM or T2DM), or rare forms of diabetes mellitus.
3. Have an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
4. Have a history of acute or chronic pancreatitis.
5. Participants with a known clinically significant gastric emptying abnormality.
6. Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy.
7. Have a history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the Investigator, may preclude the participant from following and completing the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs (Safety and tolerability) of ASC30 | Up to Day169
  A summary of AEs, SAEs and other non-serious adverse events

SECONDARY OUTCOMES:
Cmax of ASC30 | Up to Day169
  PK parameters of ASC30
Change From Baseline in Body Weight | Up to Day169
  Change From Baseline in Body Weight

CONTACTS AND LOCATIONS:
Locations (1):
- Ascletis clinical site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No